CLINICAL TRIAL: NCT05507060
Title: Evaluation of the Efficacy of Different Nebulization Techniques in Acute Exacerbation of Chronic Obstructive Pulmonary Disease Patients, Randomized, Single-blind, Clinical Trial
Brief Title: Evaluation of the Efficacy of Different Nebulization Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Erdem Cevik, Associate Prof., Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Ecevik1
Record Dates: First submitted 2022-08-05; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: COPD Exacerbation
Keywords: COPD; nebulizers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The measurements will be recorded in the patient file and the groups will be coded so that the researcher evaluating the data will be blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vibrating MESH nebulizer (Active Comparator): Medication will be applied with Vibrating MESH nebulizer
  Interventions: Device: Vibrating MESH nebulizer (Aerogen Ultra)
- Jet nebulizers (Active Comparator): Medication will be applied with Jet nebulizers
  Interventions: Device: Jet nebulizers (Philips Respironics)

INTERVENTIONS:
Device: Vibrating MESH nebulizer (Aerogen Ultra) — Medication will be applied with Vibrating MESH nebulizer
  Arms: Vibrating MESH nebulizer
Device: Jet nebulizers (Philips Respironics) — Medication will be applied with Jet nebulizers
  Arms: Jet nebulizers

SUMMARY:
COPD is the 3rd most common cause of death in the world, and the most common places of admission in our country with exacerbation of COPD are emergency services. β-2 agonists and/or short-acting anticholinergic drugs use is recommended in patients with COPD Salbutamol is known to cause significant improvement in dyspnea, quality of life and FEV1 in patients with COPD. Various techniques are used to administer drugs, one of which is the nebulization technique and is frequently used in emergency departments. There are limited clinical studies comparing different nebulization techniques, and the aim of this study is to compare the efficacy of Vibrating MESH nebulizer versus Jet nebulizers in a COPD exacerbation patient.

Patients who applied to the Emergency Department of Sultan Abdulhamid Han Training and Research Hospital with the complaint of shortness of breath and were diagnosed with COPD exacerbation according to the Gold Guidelines and to be treated with nebulization will be included in the study. Patients who agreed to participate in the study will be divided into two groups and assigned sequentially according to the simple randomization schedule.

Medication will be applied to one group with Jet nebulizers (Philips Respironics) and to the other group with Vibrating MESH nebulizer (Aerogen Ultra). Vital signs, IPI, spirometric measurements (FEV 1, FVC, FEV1 / FVC, FEF 50, FEF 2575), and dyspnea VAS score will be recorded at admission and re-measured after 1hour of treatment . In addition, single dose nebulization time will be measured and patient satisfaction will be measured with a 5-linkert scale. Demographic data will be recorded. The measurements will be recorded in the patient file and the groups will be coded so that the researcher evaluating the data will be blinded to the groups. The patient could not be blinded because of the different shape of devices.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of COPD according to GOLD guidline,
* Being over 18 years old,
* Being able to read and to understand the spoken language and give consent.

Exclusion Criteria:

* Patients who need NIMW or intubation.
* Covid 19 or suspected patients
* cognitive disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
change of spirometric measurement | Change from pretreatment spirometric measurements at first hour.
  Change of FEV 1%, FVC %, FEV1 / FVC %, FEF 50 %, FEF 2575 %
Change of Integrated pulmonary index( IPI) | Change from pretreatment IPI at first hour.
  IPI will measured by Capnostream™ 35 Portable Respiratory Monitor. The device can give single digit, 1-10. 10 is normal and 1-2 is need immediately intervention
VAS score change of dyspnea | Change from pretreatment VAS score at first hour.
  0 is no dyspnea and 10 is the biggest dyspnea attacks

SECONDARY OUTCOMES:
nebulization time | Measured with each nebulization treatment at first hour
  time from start to end of nebulization treatment will measured in minutes
patient satisfaction | Measured after each nebulization application at first hour.
  Satisfaction of nebulization treatment ( 5 Lincert scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdulhamid Han Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol will be shared but Our clinical datas' are not available for sharig considering ethical problems.

REFERENCES:
- [Background] Ashraf S, McPeck M, Cuccia AD, Smaldone GC. Comparison of Vibrating Mesh, Jet, and Breath-Enhanced Nebulizers During Mechanical Ventilation. Respir Care. 2020 Oct;65(10):1419-1426. doi: 10.4187/respcare.07639. Epub 2020 Jul 21. PMID 32694180
- [Background] Dogan NO, Varol Y, Kokturk N, Aksay E, Alpaydin AO, Corbacioglu SK, Aksel G, Baha A, Akoglu H, Karahan S, Sen E, Ergan B, Bayram B, Yilmaz S, Gurgun A, Polatli M. 2021 Guideline for the Management of COPD Exacerbations: Emergency Medicine Association of Turkey (EMAT) / Turkish Thoracic Society (TTS) Clinical Practice Guideline Task Force. Turk J Emerg Med. 2021 Oct 29;21(4):137-176. doi: 10.4103/2452-2473.329630. eCollection 2021 Oct-Dec. PMID 34849428
- [Background] Dailey PA, Shockley CM. Review of aerosol delivery in the emergency department. Ann Transl Med. 2021 Apr;9(7):591. doi: 10.21037/atm-20-4724. PMID 33987289
- [Background] Gerde P, Nowenwik M, Sjoberg CO, Selg E. Adapting the Aerogen Mesh Nebulizer for Dried Aerosol Exposures Using the PreciseInhale Platform. J Aerosol Med Pulm Drug Deliv. 2020 Apr;33(2):116-126. doi: 10.1089/jamp.2019.1554. Epub 2019 Oct 15. PMID 31613690
- [Background] Sweeney L, McCloskey AP, Higgins G, Ramsey JM, Cryan SA, MacLoughlin R. Effective nebulization of interferon-gamma using a novel vibrating mesh. Respir Res. 2019 Apr 3;20(1):66. doi: 10.1186/s12931-019-1030-1. PMID 30943978
- [Background] Kocak AO, Cakir Z, Akbas I, Gur STA, Kose MZ, Can NO, Sengun E, Gemis OF. Comparison of two scores of short term serious outcome in COPD patients. Am J Emerg Med. 2020 Jun;38(6):1086-1091. doi: 10.1016/j.ajem.2019.158376. Epub 2019 Jul 27. PMID 31378412
- [Result] Watz H, Tetzlaff K, Magnussen H, Mueller A, Rodriguez-Roisin R, Wouters EFM, Vogelmeier C, Calverley PMA. Spirometric changes during exacerbations of COPD: a post hoc analysis of the WISDOM trial. Respir Res. 2018 Dec 13;19(1):251. doi: 10.1186/s12931-018-0944-3. PMID 30545350
- See also: KOAH alevlenme ile acil servis'e başvuran hastalarda, spirometrik ölçümler, ciddiyet skorları ve laboratuvar parametrelerinin prognozu öngörmedeki değeri — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp